CLINICAL TRIAL: NCT03663751
Title: Pre-emptive Therapy With Low-dose Decitabine for Patients With Decreased Donor Chimerism After Allogeneic Stem Cell Transplantation
Brief Title: Low-dose Decitabine for the Treatment of Decreased Donor Chimerism After Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, BMT program, Deputy director, Department of Hematology, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-BMT-2018-1
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Response Rate
Keywords: donor chimerism,; decitabine,; allo-HSCT
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The peripheral and bone marrow T cell and mono nucleated cell chimerism will be closely followed-up. In case of decreasing donor chimerism, patients will receive low-dose decitabine with 5mg/m2 daily for 5 days every 6-8 weeks until the chimerism recovered to full donor type (>98%).
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — low-dose decitabine: 5mg/m2 daily for 5 days
  Other Names: LD-DAC

SUMMARY:
Decreasing donor chimerism is considered as an early sign of graft failure or relapse in patients undergoing allogeneic stem cell transplantation. The treatment option included tapering or stop of immunosuppression and or donor lymphocyte infusion (DLI) which may restore a full donor chimerism but subsequent graft versus host disease (GVHD) is the major complications. In this single arm prospective study, the investigator evaluate the effect and safety of low-dose decitabine alone or with DLI in patients with decreased donor chimerism after allo-HSCT.

DETAILED DESCRIPTION:
Decreasing donor chimerism is considered as an early sign of graft failure or relapse in patients undergoing allogeneic stem cell transplantation. The treatment option included tapering or stop of immunosuppression and or donor lymphocyte infusion (DLI) which may restore a full donor chimerism but subsequent GVHD is the major complications. In this single arm prospective study, the investigator plan to evaluate the effect and safety of low-dose decitabine treatment alone in patients with decreased donor chimerism after allo-HSCT. The investigators expect an overall response rate of 80% without serious toxicity such as grade III-IV aGVHD, ext cGVHD and lethal infection event associated with low-dose decitabine (LD-DAC) treatment. In case of donor chimerism decreasing, 5-day low-dose decitabine (5mg/m2) will given every 6 to 8 weeks until full donor chimerism is achieved (>98%). Fast withdraw of immuno-suppression or stop of immunosupression is not carried out in the study.

ELIGIBILITY:
Inclusion Criteria:

* all patients after allogeneic stem cell transplantation
* decreasing of donor chimerism to less than 97%
* providing inform consent

Exclusion Criteria:

* patients with documented relapse disease
* patients with documented positive MRD+ (>0.1% via flowcytometry or PCR)
* patients with active infection or grade III-IV GVHD

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Complete response rate | 6 months after initiation of treatment
  Documentation >98% donor chimerism of T cells or mononuclear cell in either peripheral blood or bone marrow

SECONDARY OUTCOMES:
relapse rate | 12 months after initiation of treatment
  Documentation of blast in bone marrow >5%
engraftment failure | 12 months after initiation of treatment
  Documentation of pancytopenia with donor chimerism <5%
survival rate | 12 months after initiation of treatment
  event counted as death due to any cause
incidence of grade III-IV aGVHD | 12 months after initiation of treatment
  event counted as documentation of new onset or aggravation of pre-existing aGVHD into grade III-IV
incidence of moderate to severe chronic GVHD | 12 months after initiation of treatment
  event counted as documentation of moderate to severe chronic GVHD
Overall response | 6 months after initiation of treatment
  Documentation of complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Jiong HU, Principal Investigator — Department of Hematology, Rui jin Hospital
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No